CLINICAL TRIAL: NCT03558828
Title: Testing Adaptive Interventions to Improve Physical Activity for Sedentary Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Illinois at Chicago (Other); Michigan State University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 17053108-IRB01; 5R01NR017635-04 (NIH); NCT03558828 (Registry Identifier: clinicaltrials.gov); DUNS: 068610245 (Other: Rush University Medical Center); UEI: C155UU2TXCP3 (Other: Rush University Medical Center); EIN: 1362174823A1 (Other: Rush University Medical Center)
Record Dates: First submitted 2018-04-23; First posted 2018-06-15 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Physical Activity
Keywords: physical activity; women; sedentary; accelerometer; text message; group meeting; personal call; workplace; cost-effectiveness; Sequential Multiple Assignment Randomized Trial; adaptive intervention; Actigraph; Fitbit; iCardia
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A Sequential Multiple Assignment Randomized Trial (SMART) design is used for this study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Step1: Initial Treatment (Experimental): Participants will be randomly assigned to one of the two initial treatment components: a) enhanced physical activity monitor only (physical activity monitor with goal setting and a physical activity prescription) treatment, or b) enhanced physical activity monitor+ motivational text messaging treatment for 8 weeks (early adoption phase). All participants will be given a physical activity step goal The initial treatment time period is from Weeks 1-8.
  Interventions: Behavioral: Step 1: PA Monitor; Behavioral: Step 1: PA Monitor + Text
- Step 2: Augmented Treatment (Experimental): At Week 8, it will be determined if a women has met her physical activity step goal. If she has, then she will be classified as a responder, and will continue with the same initial treatment component for weeks 9-34 (later adoption).
  If a woman has not met her physical activity step goal she will be classified as a non-responder. In addition to the initial treatment component non-responders to initial treatments will be randomly assigned to one of two augmented treatment components: a) personal calls, or b) group meetings for Weeks 9-34 (later adoption phase).
  Interventions: Behavioral: Step 2: PA Monitor with Calls; Behavioral: Step 2: PA Monitor with Meetings; Behavioral: Step 2: PA Monitor + Texts with Calls; Behavioral: Step 2: PA Monitor + Texts with Meetings
- Step 3: Maintenance (Experimental): At Weeks 35-50 (maintenance phase) all participants in the study return to an enhanced physical activity monitor only treatment component.
  Interventions: Behavioral: Step 3: PA Monitor

INTERVENTIONS:
Behavioral: Step 1: PA Monitor — The participant will receive an enhanced physical activity monitor treatment for weeks 1-8, which includes goal setting with a physical activity prescription, and self-monitoring with a physical activity monitor.
  Arms: Step1: Initial Treatment
Behavioral: Step 1: PA Monitor + Text — The participant will receive an enhanced physical activity monitor treatment for weeks 1-8, which includes goal setting with a physical activity prescription, and self-monitoring with a physical activity monitor.
  In addition, these participants will receive motivational text messages. For participants who remain less than halfway to their daily step goal by a designated daily time, a motivational text message with a strategy to overcome barriers will be sent.
  Arms: Step1: Initial Treatment
Behavioral: Step 2: PA Monitor with Calls — Nonresponders to the enhanced physical activity monitor, will receive an augmented treatment.
  The participant will continue to receive an enhanced physical activity monitor treatment for weeks 9-34.
  In addition they will receive ten brief motivational telephone calls, made by an interventionist, every two to three weeks during weeks 9-34.
  Arms: Step 2: Augmented Treatment
Behavioral: Step 2: PA Monitor with Meetings — Nonresponders to the enhanced physical activity monitor, will receive an augmented treatment.
  The participant will continue to receive an enhanced physical activity monitor treatment for weeks 9-34.
  In addition, the participant will take part in five 45-minute group meetings held every four to six weeks during Weeks 9-34.
  Arms: Step 2: Augmented Treatment
Behavioral: Step 2: PA Monitor + Texts with Calls — Nonresponders to the enhanced physical activity monitor plus text messaging, will receive an augmented treatment.
  The participant will continue to receive an enhanced physical activity monitor treatment for weeks 9-34.
  In addition, these participants will continue to receive motivational text messages. For participants who remain less than halfway to their daily step goal by a designated daily time, a motivational text message with a strategy to overcome barriers will be sent.
  In addition they will receive ten brief motivational telephone calls, made by an interventionist, every two to three weeks during weeks 9-34.
  Arms: Step 2: Augmented Treatment
Behavioral: Step 2: PA Monitor + Texts with Meetings — Nonresponders to the enhanced physical activity monitor plus text messaging, will receive an augmented treatment.
  The participant will continue to receive an enhanced physical activity monitor treatment for weeks 9-34.
  In addition, these participants will continue to receive motivational text messages. For participants who remain less than halfway to their daily step goal by a designated daily time, a motivational text message with a strategy to overcome barriers will be sent.
  In addition, the participant will take part in five 45-minute group meetings held every four to six weeks during Weeks 9-34.
  Arms: Step 2: Augmented Treatment
Behavioral: Step 3: PA Monitor — During Weeks 35-50, all women will receive enhanced physical activity monitors only.
  Arms: Step 3: Maintenance

SUMMARY:
This study employs a Sequential Multiple Assignment Randomized Trial (SMART) and aims to determine the most effective adaptive intervention combining four efficacious treatments (enhanced physical activity monitor, motivational text messages, motivational personal calls, group meetings) to increase physical activity and improve cardiovascular health among sedentary employed women.

DETAILED DESCRIPTION:
The long-term goal of this research program is to develop cost-effective strategies to increase moderate- intensity physical activity among sedentary women. Fewer than half of U.S. women meet recommendations for moderate-intensity physical activity, and thereby are at increased risk for cardiovascular disease. When provided a physical activity program, between 25-60% of women either fail to adopt it or fail to adhere after six months. Physical activity health benefits are further negatively impacted by the fact that sedentary behavior at many worksites exacerbates low physical activity. Among efficacious treatments for increasing physical activity for women, four have had promising results: (1) enhanced physical activity monitor treatment (PA monitor with goal setting and a physical activity prescription); (2) motivational text messages; (3) motivational personal calls; and (4) group meetings. While each of these treatments has proven efficacy, they differ on resource use and cost, and there is heterogeneity in response. When treatments have heterogeneity of response, adaptive interventions can help close that gap. Adaptive interventions start with an initial treatment and then transition to an augmented treatment for non-responders. This study aims to determine the most effective adaptive intervention combining four efficacious treatments (enhanced physical activity monitor, motivational text messages, motivational personal calls, group meetings) to increase physical activity (step counts per day, minutes moderate/vigorous physical activity per week) and improve cardiovascular health (aerobic fitness, body composition) among sedentary employed women. The investigators will also assess treatment effects on intervention targets (physical activity benefits, physical activity barriers, physical activity self-efficacy, and social support). A Sequential Multiple Assignment Randomized Trial (SMART) design will address the following aims: 1) Among non-responders to the initial treatments (enhanced physical activity monitor and enhanced physical activity monitor+ motivational text messages), compare the two augmented treatments (motivational personal calls and group meetings); 2a) Compare the two initial treatments and; 2b) Compare the four adaptive interventions embedded in the SMART on physical activity and cardiovascular health; 3) Identify mediators and moderators of the initial and augmented treatments on physical activity and cardiovascular health; 4) Compare the cost-effectiveness of the four adaptive interventions from the societal perspective which includes both program costs and participant costs. The investigators will recruit 312 sedentary women, aged 18 to 70, who are employed at a large urban academic medical center. Data will be collected on physical activity (self- report, device), cardiovascular health, physical activity benefits, physical activity barriers, physical activity self-efficacy, social support, and program and participant costs. Data will be collected at baseline, weeks 9-10 (when response to initial treatment is assessed), weeks 35-36, and weeks 51-52. The investigators expect to identify an optimal adaptive intervention for improving physical activity and cardiovascular health that minimizes costs and burden to women who respond to less intensive treatments, while maximizing benefits for those who need a more intensive approach.

ELIGIBILITY:
Inclusion Criteria:

* Female employee at study site
* Aged 18 to 70
* Able to speak/read English
* Owns a smartphone with text messaging capability
* Willing to receive text messages at the proposed pace
* We will include participants who have Type 1 diabetes, or Type 2 diabetes with an A1C ≥ 9.0%, or have an A1C of ≥ 6.5% without a prior diabetes diagnosis, only if they have been given clearance by their health care provider
* Without a disability that inhibits walking as determined by the PAR-Q & You (Physical Activity Readiness Questionnaire)

Exclusion Criteria

* Major signs/symptoms of pulmonary or cardiovascular disease
* Systolic BP ≥ 160 and/or diastolic BP ≥ 100
* Sufficiently or overly active, as determined by a physical activity monitor worn for one week, indicating averaging ≥ 7,500 steps per day ("somewhat active")

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 301 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Buchholz, PhD, Principal Investigator — Michigan State University, College of Nursing
Locations (1):
- Rush University College of Nursing, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchholz SW, Ingram D, Wilbur J, Fogg L, Sandi G, Moss A, Ocampo EV. Bilingual Text4Walking Food Service Employee Intervention Pilot Study. JMIR Mhealth Uhealth. 2016 Jun 1;4(2):e68. doi: 10.2196/mhealth.5328. PMID 27251878
- [Background] Wilbur J, Miller AM, Fogg L, McDevitt J, Castro CM, Schoeny ME, Buchholz SW, Braun LT, Ingram DM, Volgman AS, Dancy BL. Randomized Clinical Trial of the Women's Lifestyle Physical Activity Program for African-American Women: 24- and 48-Week Outcomes. Am J Health Promot. 2016 May;30(5):335-45. doi: 10.1177/0890117116646342. PMID 27404642
- [Background] Buchholz SW, Wilbur J, Halloway S, Schoeny M, Johnson T, Vispute S, Kitsiou S. Study protocol for a sequential multiple assignment randomized trial (SMART) to improve physical activity in employed women. Contemp Clin Trials. 2020 Feb;89:105921. doi: 10.1016/j.cct.2019.105921. Epub 2019 Dec 30. PMID 31899371
- [Background] Daniel M, Buchholz SW, Schoeny M, Halloway S, Kitsiou S, Johnson T, Vispute S, Kapp M, Wilbur J. Effects of the COVID-19 pandemic on recruitment for the working women walking program. Res Nurs Health. 2022 Oct;45(5):559-568. doi: 10.1002/nur.22258. Epub 2022 Sep 12. PMID 36093873
- [Background] Buchholz SW, Daniel M, Kitsiou S, Schoeny ME, Halloway S, Johnson TJ, Vispute S, Wilbur J. Working Women Walking Program: A Sequential Multiple Assignment Randomized Trial. J Phys Act Health. 2025 May 6;22(7):778-792. doi: 10.1123/jpah.2024-0790. Print 2025 Jul 1. PMID 40328439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Response to reviewer's comment #2- Each arm includes a specific title and time period. For Column #7 during the maintenance period, a total of 301 participants were analyzed. If we were to include "301" again in this column, the total would add up to 602, which would count the same participants twice. To avoid the double-counting and to keep the total participant number as 301, I've added column #7 but entered n as 0 in the maintenance period column.
  Comment #3. Response: footnote removed
Pre-assignment Details: Excluded: 453
  * Unable to be reached: 163
  * Not Interested: 193
  * Ineligible: 97
  * failed phone screening: 14
  * failed health screening: 33
  * failed physical activity screening: 50
Groups:
- Enhanced Physical Activity Monitor Only: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor only" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps.
  Step 2: Responder Treatment (weeks 9-34)- responders to "Enhanced Physical Activity Monitor only" treatment continued with this assigned treatment.
  Step 3: Maintenance (weeks 35-50)- responders to "Enhanced Physical Activity Monitor only" treatment continued with this assigned treatment.
- Enhanced Physical Activity Monitor+ Motivational Text Messages: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Responder Treatment (weeks 9-34)- responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment.
  Step 3: Maintenance (weeks 35-50)- responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only .
- Enhanced Physical Activity Monitor Only+ Personal Calls: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor only" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with Enhanced Physical Activity Monitor plus were randomized to receive Personal Calls.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with "Enhanced Physical Activity Monitor" only.
- Enhanced Physical Activity Monitor Only+ Group Meetings: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor only" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with Enhanced Physical Activity Monitor plus were randomized to participate in Group Meetings.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with "Enhanced Physical Activity Monitor" only.
- Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment plus were randomized to receive Personal Calls.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only .
- Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment plus were randomized to participate in Group Meetings.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only .
Period: Overall Study
Arm/Group | Enhanced Physical Activity Monitor Only | Enhanced Physical Activity Monitor+ Motivational Text Messages | Enhanced Physical Activity Monitor Only+ Personal Calls | Enhanced Physical Activity Monitor Only+ Group Meetings | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings
Started | 76 | 81 | 38 | 35 | 35 | 36
Completed | 71 | 77 | 35 | 30 | 33 | 33
Not Completed | 5 | 4 | 3 | 5 | 2 | 3
Not completed — Lost to Follow-up | 4 | 3 | 3 | 5 | 2 | 3
Not completed — dropped before the intervention | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are available for N=301 participants in Step 1 only (Weeks 1-8) as all 301 participants progressed to Steps 2 and 3.
Groups:
- Step1: Initial Treatment (Weeks 1-8) Enhanced Physical Activity Monitor Only: Step1: Initial Treatment (weeks 1-8) enhanced physical activity monitor only: In this group, participants were randomly assigned to an enhanced physical activity monitor only, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps. For baseline characteristics, this step includes both responders and non-responders from the physical activity monitor-only treatment group.
- Step1: Initial Treatment (Weeks 1-8) Enhanced Physical Activity Monitor + Text Messages: Step1: Initial Treatment (weeks 1-8) enhanced physical activity monitor +motivational text messaging: In this group, participants were randomly assigned to an enhanced physical activity monitor (Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps) + text messages. For baseline characteristics, this step includes both responders and non-responders from the physical activity monitor + text messages treatment group.
- Total: Total of all reporting groups
Arm/Group | Step1: Initial Treatment (Weeks 1-8) Enhanced Physical Activity Monitor Only | Step1: Initial Treatment (Weeks 1-8) Enhanced Physical Activity Monitor + Text Messages | Total
Number analyzed (Participants) | 149 | 152 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 149 | 152 | 301
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (11.6) | 46.1 (11.2) | 45.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 152 | 301
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 16 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 44 | 48 | 92
  White | 78 | 74 | 152
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 14 | 34
Region of Enrollment [Number; unit: participants]
  United States | 149 | 152 | 301
Average daily steps [Mean (Full Range); unit: Number of steps (M, 95% CI)] — Average daily steps reported as M (95% CI). However, M and "full range" selected since there is no option to select "95% CI".
  Number of steps (M, 95% CI) | 4913.95 [4588 to 5228] | 5082.05 [4736 to 5394] | 4998 [4588 to 5394]
Average daily minutes of moderate/vigorous PA (MVPA) [Mean (Full Range); unit: Number pf MVPA minutes/day (M, 95% CI)] — Average MVPA minutes/day are reported as M (95%) However, M and "full range" selected since there is no option to select "95% CI".
  Number pf MVPA minutes/day (M, 95% CI) | 13.5 [11.8 to 15.2] | 13.7 [11.5 to 15.8] | 13.6 [11.5 to 15.8]

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity-Steps
Description: Physical activity-Steps: Average daily steps were measured with ActiGraph worn on the right hip during waking hours for one week.
Time Frame: Baseline plus change is being assessed after 8 weeks, 34 weeks, and 50 weeks for steps.
Population: Total N=301 participants were analyzed.
Measure: Mean (95% Confidence Interval); unit: Number of steps/day
Groups:
- Enhanced Physical Activity Monitor+ Motivational Text Messages: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Responder Treatment (weeks 9-34)- responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment.
  Step 3: Maintenance (weeks 35-50)- responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only.
- Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment plus were randomized to receive Personal Calls.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only.
Arm/Group | Enhanced Physical Activity Monitor Only | Enhanced Physical Activity Monitor+ Motivational Text Messages | Enhanced Physical Activity Monitor Only+ Personal Calls | Enhanced Physical Activity Monitor Only+ Group Meetings | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings
Number analyzed (Participants) | 76 | 81 | 38 | 35 | 35 | 36
Number of steps/day | 5637.2 [5215 to 6045] | 5863.3 [5443 to 6275] | 5603.9 [5164 to 6044] | 5631.6 [5194 to 6070] | 5636.7 [5214 to 6060] | 5322.0 [4892 to 5752]
Statistical Analysis 1: Comparison: Enhanced Physical Activity Monitor Only vs Enhanced Physical Activity Monitor+ Motivational Text Messages vs Enhanced Physical Activity Monitor Only+ Personal Calls vs Enhanced Physical Activity Monitor Only+ Group Meetings vs Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls vs Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings; Test type: Other — A power analysis based on the study's primary aim (impact of augmented treatments on non-responders) was conducted. An estimated effect size of d=0.41 for the difference between the two augmented treatments was used. With a 2-tailed alpha of 0.05, a pre-post correlation of r=0.60, and a sample size of 188 non-responders, an estimated 80% power was obtained. Assuming 67% non-response to the initial treatments and 10% attrition, the final target sample size was N=312; GEEs — All analyses employed an intent-to-treat approach using a two-tailed alpha of 0.05 with no adjustment for multiple tests; Effect size estimates = .41 — Effect size estimates (Cohen's d) for all analyses were created by using the relevant slope (i.e., change) effect as the numerator and the baseline standard deviation of the dependent variable as the denominator; The longitudinal trajectories using generalized estimating equations (GEEs) were estimated. Cases for responders are duplicated and weighted based on the inverse probability of being assigned to a particular adaptive intervention (i.e., responders have a ½ probability of assignment to a specific adaptive intervention, and non-responders have a ¼ probability). Only the Phase 1 (baseline to 8 weeks) treatment condition x time interaction was included because it preceded the randomization to Phase 2 (weeks 9-34) treatment conditions. Planned contrasts were used to test specific hypotheses. Effect size estimates for all analyses were created by using the relevant slope effect as the numerator and the baseline standard deviation of the dependent variable as the denominator. All analyses employed an intent-to-treat approach using a two-tailed alpha of 0.05 with no adjustment for multiple tests

2. Primary Outcome: Physical Activity- Moderate to Vigorous Physical Activity (MVPA)
Description: Average daily minutes of Moderate to Vigorous Physical Activity (MVPA) were measured with ActiGraph worn on the right hip during waking hours for one week.
Time Frame: Baseline plus change is being assessed after 8 weeks, 34 weeks, and 50 weeks for MVPA.
Population: Total N=301 participants were analyzed.
Measure: Mean (95% Confidence Interval); unit: Number of MVPA minutes/day
Groups:
- Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings: Step 1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment plus were randomized to participate in Group Meetings.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only.
Arm/Group | Enhanced Physical Activity Monitor Only | Enhanced Physical Activity Monitor+ Motivational Text Messages | Enhanced Physical Activity Monitor Only+ Personal Calls | Enhanced Physical Activity Monitor Only+ Group Meetings | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings
Number analyzed (Participants) | 76 | 81 | 38 | 35 | 35 | 36
Number of MVPA minutes/day | 17.4 [14.9 to 19.7] | 18.0 [15.2 to 21.1] | 18.8 [15.5 to 22.2] | 17.9 [14.8 to 21.0] | 18.6 [15.7 to 21.5] | 17.7 [14.1 to 21.3]
Statistical Analysis 1: Comparison: Enhanced Physical Activity Monitor Only vs Enhanced Physical Activity Monitor+ Motivational Text Messages vs Enhanced Physical Activity Monitor Only+ Personal Calls vs Enhanced Physical Activity Monitor Only+ Group Meetings vs Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls vs Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings; Test type: Other — [test comment as in outcome 1, analysis 1]; GEEs — [p-value comment as in outcome 1, analysis 1]; Effect size estimates = .41 — Effect size estimates for all analyses were created by using the relevant slope (i.e., change) effect as the numerator and the baseline standard deviation of the dependent variable as the denominator. An estimated effect size of d=0.41 was used; There were time slope terms for Phase 1 (baseline to 8-week assessment), Phase 2 (9-weeks to 34-week assessment), and Phase 3 (maintenance from 35-weeks to 50-week assessment). Also, there were interactions of condition and time slopes. For Phase 1, only the Phase 1 treatment condition x time interaction was included because it preceded the randomization to Phase 2 treatment conditions. Supplementary analyses were conducted to compare the trajectories of responders versus non-responders to the Phase 1 treatment. Effect size estimates for all analyses were created by using the relevant slope (i.e., change) effect as the numerator and the baseline standard deviation of the dependent variable as the denominator. The resulting effect size is equivalent to a Cohen's d, representing mean change (or difference in change) in standard deviation units. All analyses employed an intent-to-treat approach using a two-tailed alpha of 0.05 with no adjustment for multiple tests

3. Secondary Outcome: Cardiovascular Health (1)
Description: Aerobic fitness: participants step in place to a predesignated height for 2 minutes and the average number of steps taken in 2 minutes are counted.
Time Frame: Baseline plus change is being assessed after 8 weeks, 34 weeks, and 50 weeks for aerobic fitness.
Population: Total N=301 participants were analyzed.
Measure: Mean (95% Confidence Interval); unit: Number of steps/2 minutes
Groups:
- Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls: Step2: Augmented Treatment (weeks 9-34) enhanced physical activity monitor + text messages + personal calls: In this group, participants who were non-responders to the enhanced physical activity monitor + text messages in step 1, continued with enhanced PA monitor + text messages + were randomized to receive personal calls.Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment plus were randomized to receive Personal Calls.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only.
Arm/Group | Enhanced Physical Activity Monitor Only | Enhanced Physical Activity Monitor+ Motivational Text Messages | Enhanced Physical Activity Monitor Only+ Personal Calls | Enhanced Physical Activity Monitor Only+ Group Meetings | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings
Number analyzed (Participants) | 76 | 81 | 38 | 35 | 35 | 36
Number of steps/2 minutes | 85.7 [81.5 to 90.1] | 87.1 [82.2 to 92.2] | 86.3 [81.2 to 91.4] | 89.9 [85.2 to 94.7] | 86 [81.4 to 90.6] | 88.7 [83.9 to 93.5]

4. Secondary Outcome: Cardiovascular Health (2)
Description: Body composition: Average BMI (weight measured in pounds; height measured in inches) was measured utilizing BMI calculation formula: BMI = Weight (kg) / Height (m)²
Time Frame: Baseline plus change is being assessed after 8 weeks, 34 weeks, and 50 weeks for BMI.
Population: Total N=301 participants were analyzed.
Measure: Mean (95% Confidence Interval); unit: weight (pounds)/height (Inches)^2x703
Groups:
- Enhanced Physical Activity Monitor Only+Personal Calls: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor only" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with Enhanced Physical Activity Monitor plus were randomized to receive Personal Calls.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with "Enhanced Physical Activity Monitor" only.
Arm/Group | Enhanced Physical Activity Monitor Only | Enhanced Physical Activity Monitor+ Motivational Text Messages | Enhanced Physical Activity Monitor Only+Personal Calls | Enhanced Physical Activity Monitor Only+ Group Meetings | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings
Number analyzed (Participants) | 76 | 81 | 38 | 35 | 35 | 36
weight (pounds)/height (Inches)^2x703 | 31.8 [30.4 to 33.2] | 32.4 [30.8 to 34.2] | 31.3 [29.8 to 32.8] | 31.6 [30.1 to 33.1] | 32.2 [30.6 to 33.9] | 32.1 [30.5 to 33.8]

5. Secondary Outcome: Cardiovascular Health (3)
Description: Body composition: Average waist circumference was measured in inches.
Time Frame: Baseline plus change is being assessed after 8 weeks, 34 weeks, and 50 weeks for waist measurement.
Population: Total N=301 participants were analyzed.
Measure: Mean (95% Confidence Interval); unit: Inches
Groups:
- Enhanced Physical Activity Monitor Only+ Personal Calls Activity Monitor Only + Personal Calls: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor only" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with Enhanced Physical Activity Monitor plus were randomized to receive Personal Calls.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor only" treatment continued with "Enhanced Physical Activity Monitor" only.
Arm/Group | Enhanced Physical Activity Monitor Only | Enhanced Physical Activity Monitor+ Motivational Text Messages | Enhanced Physical Activity Monitor Only+ Personal Calls Activity Monitor Only + Personal Calls | Enhanced Physical Activity Monitor Only+ Group Meetings | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings
Number analyzed (Participants) | 76 | 81 | 38 | 35 | 35 | 36
Inches | 38.1 [36.9 to 39.4] | 38.7 [36.9 to 40.0] | 38.4 [37.1 to 39.7] | 39 [37.8 to 40.2] | 39.8 [38.4 to 41.2] | 38.7 [37.4 to 40.0]

ADVERSE EVENTS:
Time Frame: Monitored during Step 1: initial treatment period (weeks 1-8), Step 2: augmented treatment period (weeks 9-34), and Step 3: Maintenance period (weeks 35-50)
Description: Included all participants (N=301) in initial treatment period (weeks 1-8), augmented treatment period (weeks 9-34), and Maintenance period (weeks 35-50).
Groups:
- Enhanced Physical Activity Monitor Only+ Group Meetings; Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls: Step1: Initial Treatment (weeks 1-8)- participants were randomly assigned to an "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment, which included Fitbit with goal setting, a physical activity prescription, and self-monitoring of daily steps + Text Messages.
  Step 2: Non-responder Treatment (weeks 9-34)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with this assigned treatment plus were randomized to receive Personal Calls.
  Step 3: Maintenance (weeks 35-50)- non-responders to "Enhanced Physical Activity Monitor + Motivational Text Messages" treatment continued with "Enhanced Physical Activity Monitor" only.
Arm/Group | Enhanced Physical Activity Monitor Only | Enhanced Physical Activity Monitor+ Motivational Text Messages | Enhanced Physical Activity Monitor Only+ Personal Calls | Enhanced Physical Activity Monitor Only+ Group Meetings | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/81 | 0/38 | 0/35 | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/81 | 0/38 | 0/35 | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 3/76 | 0/81 | 0/38 | 0/35 | 0/35 | 0/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Physical Activity Monitor Only (N=76) | Enhanced Physical Activity Monitor+ Motivational Text Messages (N=81) | Enhanced Physical Activity Monitor Only+ Personal Calls (N=38) | Enhanced Physical Activity Monitor Only+ Group Meetings (N=35) | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Personal Calls (N=35) | Enhanced Physical Activity Monitor+ Motivational Text Messages+ Group Meetings (N=36)
Elevated blood pressure (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 3 events of elevated blood pressure (3 different participants). All 3 reported following up with primary care providers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT03558828/Prot_007.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT03558828/SAP_000.pdf
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03558828/ICF_008.pdf